CLINICAL TRIAL: NCT07342114
Title: A Phase I Dose-Escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of RO7875913 in Healthy Volunteers
Brief Title: A Dose-Escalation Study of RO7875913 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GO46451
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RO7875913 (Experimental): Participants will receive RO7875913.
  Interventions: Drug: RO7875913
- Placebo (Placebo Comparator): Participants will receive Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7875913 — Participants will receive RO7875913 as per the schedule described in the protocol.
  Arms: RO7875913
Drug: Placebo — Participants will receive placebo as per the schedule described in the protocol.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and pharmacodynamics of RO7875913 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to adhere to the contraception requirements
* Body weight > 40 kilogram (kg) with a body mass index of 18-30 kg per meter square (kg/m^2)

Exclusion Criteria:

* Positive test result for hepatitis B surface antigen, hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody screen
* History of any malignancy
* Major surgical procedure within 28 days prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History or clinical manifestations of significant metabolic, hepatic, renal, pulmonary, cardiovascular, hematologic, gastrointestinal, urologic, neurologic, or psychiatric disorders
* Known allergy or hypersensitivity to any component of the RO7875913 formulation
* Treatment with investigational biologic therapy (or blinded comparator) within 90 days or 5 drug elimination half-lives, whichever is longer, prior to initiation of study drug
* Treatment with investigational non-biologic therapy (or blinded comparator) within 28 days or 5 drug elimination half-lives, whichever is longer, prior to initiation of study drug
* Treatment with any immunosuppressive medication within 28 days or 5 drug elimination half-lives, whichever is longer, prior to initiation of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-03 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to approximately 3 months

SECONDARY OUTCOMES:
Serum concentration of RO7875913 | Up to Day 76
Percentage of Participants with Anti-Drug Antibodies (ADAs) to RO7875913 at Baseline and with ADAs to RO7875913 During the Treatment Period | Baseline, Up to Day 76
Recommended Phase II Dose (RP2D) of RO7875913 | Up to approximately 3 months
Observed Value of Pharmacodynamic Markers | Baseline, up to approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.

IPD SHARING:
Plan to Share IPD: No